CLINICAL TRIAL: NCT02788500
Title: The Sports-Related Injuries and Illnesses in Para-sport Study (SRIIPS): A Prospective Longitudinal Study
Brief Title: The Sports-Related Injuries and Illnesses in Para-sport Study (SRIIPS)
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Jan Lexell, Professor, Lund University
Other Study IDs: P2016-0069
Record Dates: First submitted 2016-05-22; First posted 2016-06-02 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Athletic Injuries
Keywords: Epidemiology; Sports medicine; Research protocol; Athletic injuries; Sports for persons with disabilities
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Swedish para-athletes: The total population of athletes in the Swedish Paralympic program, which covers candidates for the Paralympic Summer or Winter Games, will be invited by mail to participate in the study and report their incidence of sports-related injuries and illnesses
  Interventions: Other: Incidence of sports-related injuries and illnesses

INTERVENTIONS:
Other: Incidence of sports-related injuries and illnesses — The SRIIP-study is an epidemiological cohort study aimed to prospectively collect self-report data on sports-related injuries and illnesses incidence and risk exposure during training and competition for approximately one year among Swedish para-athletes.

SUMMARY:
The overall aim of this project is to gain an in-depth understanding of the epidemiology of sports-related injuries and illnesses in parasport in order to assist the identification and development of specific injury prevention strategies adapted to parasport.

DETAILED DESCRIPTION:
The Paralympic Games is today one of the largest sport event in the world. During the last decades parasport has in many ways become elite sport, allowing people with disabilities to achieve extraordinary heights of functional capability. With the growing number of athletes there is an increased interest in athletes' health and safety, both to enhance sports performance and to prevent injuries.

Even though it is well-known that participation in sports places the athlete at risk for injuries, there are few studies covering sports-related injuries and illnesses in parasport (SRIIP). Today, some injuries and illnesses are known to be preventable. However, this requires regular monitoring of internal and external load during athletic preparation. Standardized injury surveillances have been implemented within several sports for abled-bodied athletes, but such studies do not yet exist within parasport.

In our review article (Fagher & Lexell 2014) the investigators showed that existing studies of sports-related injuries in athletes with disabilities have a variable quality and that specific disability related factors have not been examined. Further studies are therefore warranted to obtain an increased in-depth knowledge of SRIIP. With a systematic longitudinal surveillance system tailored to parasport it would be possible to observe trends and risk factors over time, and thereby have a basis for developing specific preventive measures.

The overall aim of this project is to gain an in-depth understanding of the epidemiology of SRIIP in parasport in order to assist the identification and development of specific injury prevention strategies adapted to parasport.

The specific aims are: i) to design and implement a study protocol for prospective epidemiological studies of SRIIP in parasport; ii) to prospectively estimate the annual incidence of SRIIP among Swedish Paralympic athletes; and iii) to explore risk factors and mechanisms for sustaining SRIIP based on athlete exposure in order to form the basis for moving towards safe participation in parasport.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Being a registered competitive athlete within the Swedish Paralympic Program/Organization
* Being able to communicate in Swedish and having the opportunity to every week answer a web-based questionnaire.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The total population of athletes (n=approximately 100) in the Swedish Paralympic program, which covers possbile candidates for the Paralympic Games.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2016-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Incidence of sports-related injuries and illnesses | Weekly during one year
  The athletes will be asked to self-report incidence of sports-related injuries and illnesses based on the surveillence systems developed by Jacobsson et al 2010 and Timpka 2014.

SECONDARY OUTCOMES:
Exposure of training | Weekly during one year
  The athletes will be asked to report exposure and perceived exertion of training (hours and minutes of training and rated perceived exertion (RPE) based on the RPE-scale).
Pain | Weekly during one year
  The athletes will be asked to report their perceived pain during the week on a visual analogue scale (VAS) scale.
General well-being | Weekly during one year
  The athletes will be asked to report their perceived general well-being based on questions from the Health-related quality of life questionnaire EQ-5D.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Lexell, Professor, Principal Investigator — Lund University
Locations (1):
- Rehabilitation Medicine Research group, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fagher K, Lexell J. Sports-related injuries in athletes with disabilities. Scand J Med Sci Sports. 2014 Oct;24(5):e320-31. doi: 10.1111/sms.12175. Epub 2014 Jan 15. PMID 24422719
- [Background] Jacobsson J, Timpka T, Ekberg J, Kowalski J, Nilsson S, Renstrom P. Design of a protocol for large-scale epidemiological studies in individual sports: the Swedish Athletics injury study. Br J Sports Med. 2010 Dec;44(15):1106-11. doi: 10.1136/bjsm.2009.067678. Epub 2010 May 19. PMID 20484318
- [Background] Timpka T, Alonso JM, Jacobsson J, Junge A, Branco P, Clarsen B, Kowalski J, Mountjoy M, Nilsson S, Pluim B, Renstrom P, Ronsen O, Steffen K, Edouard P. Injury and illness definitions and data collection procedures for use in epidemiological studies in Athletics (track and field): consensus statement. Br J Sports Med. 2014 Apr;48(7):483-90. doi: 10.1136/bjsports-2013-093241. PMID 24620036
- [Derived] Lexell J, Loven G, Fagher K. Incidence of sports-related concussion in elite para athletes - a 52-week prospective study. Brain Inj. 2021 Jul 3;35(8):971-977. doi: 10.1080/02699052.2021.1942551. Epub 2021 Jun 29. PMID 34185611
- [Derived] Fagher K, Jacobsson J, Dahlstrom O, Timpka T, Lexell J. An eHealth Application of Self-Reported Sports-Related Injuries and Illnesses in Paralympic Sport: Pilot Feasibility and Usability Study. JMIR Hum Factors. 2017 Nov 29;4(4):e30. doi: 10.2196/humanfactors.8117. PMID 29187343
- [Derived] Fagher K, Jacobsson J, Timpka T, Dahlstrom O, Lexell J. The Sports-Related Injuries and Illnesses in Paralympic Sport Study (SRIIPSS): a study protocol for a prospective longitudinal study. BMC Sports Sci Med Rehabil. 2016 Aug 30;8(1):28. doi: 10.1186/s13102-016-0053-x. eCollection 2016. PMID 27579170